CLINICAL TRIAL: NCT05162248
Title: Clinicopathological Outcomes of Microsatellite Instability in Colorectal Cancer
Brief Title: Microsatellite Instability in Colorectal Cancers
Acronym: MSI-CRC
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Taygun Gulsen, MD, General Surgeon, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Other Study IDs: s2021.crc
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Microsatellite Instability High; Microsatellite Instability Low; Microsatellite Instability-High
Keywords: Colorectal cancer; Prognostic factor; Microsatellite instability; Prognosis; Survival
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microsatellite instability: Immunohistochemical analysis was performed for Microsatellite Instability (MSI) status of colorectal tumors tissue.
  Interventions: Diagnostic Test: Microsatellite instability analysis

INTERVENTIONS:
Diagnostic Test: Microsatellite instability analysis — Molecular analysis for Microsatellite Instability (MSI) status was performed using immunohistochemistry (IHC). IHC now recognized as an approved method to highly precision predict MSI in colorectal cancer.

SUMMARY:
In this study, we aimed to identify the different histopathological features of tumors with microsatellite instability (MSI) compared to microsatellite stable (MSS) in patients who underwent surgery for colorectal cancer. We also planned to determine how MSI affects prognostic parameters.

DETAILED DESCRIPTION:
According to Global Cancer Statistics, higher than 1.9 million new cases of colorectal cancer (CRC) and 935,000 deaths are estimated to occur in 2020, representing about one in 10 cancer cases and deaths. Overall, it ranks third in colorectal incidence but second in mortality.

In CRC evolution, the acquisition of genomic instability is a critical point, and there are at least two different pathways in the pathogenesis of CRC: the chromosomal instability (CIN) pathway (85%) and the microsatellite instability (MSI) pathway (15%).

Microsatellite instability (MSI) is a phenotype that occurs due to a malfunction in the DNA repair mechanism and is seen in approximately 15% of colorectal cancers (CRCs). CRCs with MSI have different clinical features, such as a tendency to settle in the proximal colon, poor differentiation, and more lymphocytic infiltration in the tumor. It has been shown that CRCs with MSI have a better prognosis and respond differently to chemotherapy than CRCs with microsatellite stable (MSS).

We aimed to evaluate the different histopathological features of tumors with MSI compared to MSS in patients who underwent surgery for colorectal cancer. We also planned to determine how MSI affects prognostic parameters such as mortality rate, recurrence, disease-free survival, cancer-specific survival, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal surgery patients
* Complete follow-up information

Exclusion Criteria:

* Whose MSI status was not studied in the pathology material
* Missing follow-up information
* Colorectal resection for non-neoplastic diseases

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population of the research consists of patients undergoing colorectal surgery at the Health Sciences University Sultan 2. Abdulhamid Training and Research Hospital between March 2017 and March 2021.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Five years
  Overall survival is defined as the time interval from the time of primary operation to the date of all-cause death or the last follow-up.
Disease-Free Survival | Five years
  Disease-Free Survival is defined as the time interval from the time of primary operation to disease recurrence or death.

CONTACTS AND LOCATIONS:
Overall Officials: Taygun Gülşen, MD, Principal Investigator — Sultan 2. Abdulhamid Training and Research Hospital
Locations (1):
- Sultan 2. Abdulhamid Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gupta R, Sinha S, Paul RN. The impact of microsatellite stability status in colorectal cancer. Curr Probl Cancer. 2018 Nov;42(6):548-559. doi: 10.1016/j.currproblcancer.2018.06.010. Epub 2018 Jul 18. PMID 30119911
- [Background] Boland CR, Goel A. Microsatellite instability in colorectal cancer. Gastroenterology. 2010 Jun;138(6):2073-2087.e3. doi: 10.1053/j.gastro.2009.12.064. PMID 20420947